CLINICAL TRIAL: NCT01916941
Title: Neural Mechanisms of Change During the Treatment of Alcohol Use Disorders With Prazosin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Claire E Wilcox, MD, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1K23AA021156-01A1 (NIH)
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Active Comparator): Prazosin titrated to 16 mg daily x 6 weeks
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): Placebo X 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin
  Arms: Prazosin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study uses neurobiological measures through brain imaging, neuropsychological measures, and selfreport measures to try to understand how an effective treatment for alcoholism works. On the whole, less than 50% of people with alcoholism get better with treatment. This study will help researchers develop better treatments for alcoholism because if the investigators know why the treatments the investigators use are working, and in whom the treatments work best, then the investigators may be able to make treatment more effective by targeting treatments to individuals who would be most likely to benefit and by guiding development of more effective treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-65 meeting DSM-IV criteria for alcohol dependence in the past year;
2. seeking but not currently receiving treatment;
3. able to provide voluntary informed consent;
4. have at least 4 drinking days in the past 30 days
5. english-speaking
6. have a primary care physician or psychiatrist willing to continue prazosin if the patient tolerates it well and is finding it beneficial.

Exclusion Criteria:

1. severe neurological (e.g., head injury/stroke) conditions, Meniere's disease, narcolepsy, benign positional vertigo, heart disease or unstable angina, history of dysrhythmia/syncope, SBP<110, SBP>160, DBP>110, HR<55, HR>110, irregular heart rhythm, chronic renal or hepatic failure, pancreatitis or insulin-dependent diabetes, or other medical problems requiring immediate attention;
2. schizophrenia, schizoaffective disorder, PTSD, Bipolar I disorder, suicidal thoughts within the last month;
3. current dependence on another drug of abuse (except nicotine);
4. contraindications to MRI (e.g., pacemaker);
5. active legal problems with the potential to result in incarceration;
6. pregnancy or lactation, or child bearing age and not on birth control;
7. currently receiving treatment for alcohol dependence;
8. current use of psychoactive medications including SSRI's and other antidepressants, anti-craving medications, anxiolytics including benzodiazepines, antipsychotics, mood stabilizers or anticonvulsants;
9. history of seizures or DT's during alcohol withdrawal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Department of Psychiatry, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin: Prazosin titrated to 16 mg daily x 6 weeks
  Prazosin
- Placebo: Placebo X 6 weeks
  Placebo
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 18 | 18
Completed | 13 | 14
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 12 | 11 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Standard Alcoholic Drinks Consumed Per Week (Drinks Per Week)
Time Frame: from 2-4 weeks and from 4-6 weeks
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 18 | 18
drinks per week
  from 2-4 weeks | 13.65 (18.92) | 14.55 (17.29)
  from 4-6 weeks | 15.11 (23.66) | 11.11 (15.01)

ADVERSE EVENTS:
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/18 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin (N=18) | Placebo (N=18)
Dizziness on standing (Cardiac disorders) | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No